CLINICAL TRIAL: NCT07320742
Title: Comparison of the Effects of Fast and Slow Pranayama Techniques on Respiratory, Cardiovascular, Balance, and Psychosocial Parameters in University Students
Brief Title: Fast vs. Slow Pranayama for Breathing, Heart, Balance, and Well-Being in Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, gorkem ata, Principal Investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-4030
Record Dates: First submitted 2025-12-08; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-08

CONDITIONS: No Condition
Keywords: pranayama; pulmonary function test; breathing exercise; oxygen saturation; Stress, Psychological; postural balance
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Slow Pranayama Group (Experimental)
  Interventions: Behavioral: Slow Pranayama
- Fast Pranayama Group (Experimental)
  Interventions: Behavioral: Fast Pranayama

INTERVENTIONS:
Behavioral: Slow Pranayama — Participants will practice pranayama in a quiet room, comfortably seated (sukhasana), maintained at a comfortable temperature (24 ± 2°C). Sessions typically take place as follows:
  Participants in the Slow Pranayama Group will practice the Anuloma Viloma, Savitri, and Ujjayi breathing techniques. Slow pranayama breathing will be practiced for two minutes, with one-minute rests between each breathing technique, for a total of three cycles. Each cycle will last approximately nine minutes. Participants in both groups will rest in savasana for 10 minutes at the end of the session.
  No drugs or devices are used. The intervention is a controlled breathing exercise technique.
  Arms: Slow Pranayama Group
Behavioral: Fast Pranayama — Participants will practice pranayama in a quiet room, comfortably seated (sukhasana), maintained at a comfortable temperature (24 ± 2°C). Sessions will typically be conducted as follows:
  Participants in the Fast Pranayama Group will practice Kapalabhati, Bhastrika, and Agnisar breathing. Each breathing technique will be practiced for one minute, followed by a one-minute rest. This will be practiced for a total of four cycles. Each cycle will last approximately six minutes.
  No drugs or devices are used. The intervention is a controlled breathing exercise technique.
  Arms: Fast Pranayama Group

SUMMARY:
The goal of this clinical trial is to compare the effects of slow and rapid pranayama techniques on respiratory, cardiovascular, balance, and psychosocial parameters in healthy adults aged 18-35 years.

The main questions it aims to answer are:

Do slow and rapid pranayama techniques produce different improvements in lung volumes and peak cough flow?

Does slow pranayama lead to greater improvements in oxygen saturation and cardiovascular parameters, while rapid pranayama provides greater gains in balance and respiratory flow values?

Researchers will compare a slow pranayama group (n = 39) and a rapid pranayama group (n = 39) to determine how breathing speed influences physiological and psychosocial outcomes.

Participants will:

Be randomly assigned to one of two groups (slow or rapid pranayama).

Practice their assigned pranayama techniques for 25-30 minutes, 4 days per week for 12 weeks (one supervised, three home-based sessions).

Undergo pre- and post-intervention assessments including spirometry (FVC, FEV₁, FEF25%-75%, PEF), oxygen saturation, peak cough flow, blood pressure, heart rate, balance tests (single-leg stance, Y-Balance Test), and validated questionnaires for perceived stress, anxiety, depression, fatigue, and sleep quality.

This study aims to clarify how controlled breathing speed influences respiratory efficiency, cardiovascular regulation, postural stability, and mental well-being in young adults, contributing to evidence-based recommendations for integrating pranayama into stress-management and preventive rehabilitation programs.

ELIGIBILITY:
Inclusion Criteria:

* Between age 18-35

Exclusion Criteria:

* Subjects who have practiced yoga techniques in the last year.
* Subjects with a history of previous or current organic disease.
* Subjects who cannot practice pranayama due to physical abnormalities.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79 (Estimated)
Dates: Start 2025-08-16 (Actual); Primary Completion 2025-10-21 (Actual); Study Completion 2026-01-05 (Estimated)

PRIMARY OUTCOMES:
Forced Expiratory Flow at 25-75% of FVC (FEF25-75) | From enrollment to the end of treatment at 12 weeks
  FEF25-75 is the average flow rate during the middle half of the FVC maneuver. It is often considered a sensitive indicator of small airway function. Measurements will be carried out using the COSMED PONY FX (Italy) device, ensuring compliance with ATS/ERS standards. The values will be recorded in liters per second (L/s).

SECONDARY OUTCOMES:
Forced Vital Capacity (FVC) | From enrollment to the end of treatment at 12 weeks
  Forced Vital Capacity (FVC) represents the maximum volume of air that can be forcibly expelled from the lungs after taking the deepest possible breath. Measurements will be performed in accordance with ATS/ERS guidelines. All pulmonary function measurements will be performed using a spirometer (COSMED PONY FX®, Italy). The highest value obtained from three acceptable and repeatable maneuvers will be recorded in liters (L).
Forced Expiratory Volume in 1 Second (FEV1) | From enrollment to the end of treatment at 12 weeks
  FEV1 measures the volume of air exhaled during the first second of the FVC maneuver. It is a critical indicator of airway patency and respiratory muscle function. Data collection will be conducted using the COSMED PONY FX (Italy) device, following the ATS/ERS standardization guidelines. Results will be expressed in liters (L).
FEV1/FVC Ratio | From enrollment to the end of treatment at 12 weeks
  This parameter represents the ratio of FEV1 to FVC, which is used to differentiate between obstructive and restrictive ventilatory patterns. The measurements will be obtained using the COSMED PONY FX (Italy) spirometer, adhering to ATS/ERS guidelines. The result is expressed as a decimal ratio or percentage.
Peak Expiratory Flow (PEF) | From enrollment to the end of treatment at 12 weeks
  Peak Expiratory Flow (PEF) is the maximum flow rate achieved during a forced expiratory maneuver starting from full inspiration. It reflects the caliber of the large airways and the strength of the expiratory muscles. The measurements will be recorded using the COSMED PONY FX (Italy) spirometer according to ATS/ERS criteria, with the highest value reported in liters per second (L/s) or liters per minute (L/min).
Peak Cough Flow (PCF) | From enrollment to the end of treatment at 12 weeks.
  Peak cough flow (PCF) will be assessed using a handheld flow meter (Expirite® DL-F03). For all primary measurements, the highest value obtained from three replicates will be used in the analysis.
Oxygen Saturation | From enrollment to the end of treatment at 12 weeks
  It will be evaluated with a pulse oximeter (Freely SHO-3002) attached to the fingertip.
Blood Pressure | From enrollment to the end of treatment at 12 weeks
  Cardiovascular parameters will be measured after participants rest in a supine position for 10 minutes. Systolic and diastolic blood pressure measurements will be taken with a non-invasive OMRON M2 Intelli IT HEM-7143T1-EBK automatic blood pressure monitor (OMRON Healthcare Europe B.V., Netherlands).
Static Balance | From enrollment to the end of treatment at 12 weeks
  Static balance will be assessed using the one-leg stance test. In this test, participants will be asked to lift the foot on the tested side approximately 5 cm above the medial malleolus of the other foot while standing and maintain this position. The test will conclude when the foot touches the ground. Successful completion of the test is demonstrated by the participant's ability to maintain the position for 30 seconds. The best score from three repetitions will be recorded.
Dynamic Balance | From enrollment to the end of treatment at 12 weeks
  Dynamic balance ability will be assessed with the Y Balance Test (YDT). The YDT is a frequently used dynamic test to objectively assess lower extremity function and balance. Performance on this test is quantified as a measure of maximum reach in a specific direction or as a calculated composite score (average reach across all reach directions). During the test, participants are asked to maintain balance while reaching in the anterior, posterolateral, and posteromedial directions using their right and left feet. To calculate the test score, the average reach distance in each direction is calculated in centimeters by averaging three trials for each direction. This value is then divided by the participant's leg length and multiplied by 100 to calculate the distance in each direction as a percentage.
Anxiety | From enrollment to the end of treatment at 12 weeks
  Beck Anxiety Inventory (BAI) It is a 21-item, four-point Likert-type scale designed to measure an individual's anxiety severity over the past week. Each item is scored from 0 to 3. A total score between 8 and 15 indicates low anxiety; 16-25 indicates moderate anxiety; and 26-63 indicates high anxiety.
Depression | From enrollment to the end of treatment at 12 weeks
  Beck Depression Inventory (BDI) The BDI is a 21-item inventory; each item represents a symptom of depression. The BDI, a self-report instrument, is the most widely used depression measurement tool worldwide. Respondents rate 21 symptoms of depression on a 4-point scale ranging from 0 to 3. Therefore, total scores range from 0 to 63, with higher scores indicating greater depression severity.
Perceived Stress | From enrollment to the end of treatment at 12 weeks
  Stress level is going to evaluate with the Perceived Stress Scale (PSS), it consists of 14 items and is designed to measure the degree to which a person perceives certain life situations as stressful. Participants rate each item on a 5-point Likert-type scale ranging from "Never (0)" to "Very often (4)." Seven of the positively worded items are reverse-scored. Scores range from 0 to 56. Higher scores indicate greater perceived stress.
Fatigue Level | From enrollment to the end of treatment at 12 weeks
  The Fatigue Severity Scale (FSS), consists of nine items. For each question, the patient is asked to select a number between 1 and 7 indicating how much they agree with each statement, with 1 indicating strongly disagree and 7 indicating strongly agree. A score of 4 or higher generally indicates severe fatigue.
Sleep Quality | From enrollment to the end of treatment at 12 weeks
  Pittsburgh Sleep Quality Index (PSQI) The PSQI is a self-assessment tool that provides detailed information about sleep quality and the type and intensity of sleep disturbances over the past month. The index consists of 24 items, five of which are answered by the individual's sleep partner or roommate. The PSQI provides scores for seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, sleeping pill use, and daytime dysfunction. Each item is scored between 0 and 3. The sum of the scores for these seven components provides the PSQI score. The total PSQI score ranges from 0 to 21. A total score of 5 or less is considered to have "good" sleep quality, while a score above 5 indicates "poor" sleep quality. A PSQI score above 5 indicates that the individual has severe sleep problems in at least two different components or mild or moderate problems in more than three components. The sc

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided